CLINICAL TRIAL: NCT06299215
Title: Factors Associated With the Prognosis of Patients Admitted to for Acute Obstructive Pyelonephritis
Brief Title: Factors and Prognosis of Obstructive Pyelonephritis Patients
Acronym: PYELO-OBS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240044
Record Dates: First submitted 2024-02-09; First posted 2024-03-07 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Pyelonephritis; Prognostic
Keywords: acute kidney injury; renal remplacement therapy; hemodialysis; acute respiratory distress; hemodynamic failure
MeSH Terms: conditions — Pyelonephritis; Acute Kidney Injury; Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute obstructive pyelonephritis is a condition with a high risk of complications and may require admission to the intensive care unit.

Most of the available data on this condition comes from small, retrospective, single-centre series.

To date, no large-scale study has examined the factors associated with the prognosis of patients admitted to intensive care for acute obstructive pyelonephritis.

The aim of this study is to describe the population and prognosis of patients admitted to the intensive care unit for the management of acute obstructive pyelonephritis, and to identify factors associated with a poor prognosis in these patients.

DETAILED DESCRIPTION:
The retrospective and multicenter study consists of a retrospective and pseudonymous collection of data from medical reports of patients treated, over the period 2015-2022, in each intensive care unit agreeing to participate, .

Investigators from each participating center will be responsible for screening on all hospitalized patients over the period 2015-2022. Patients who have been hospitalized for the management of acute obstructive pyelonephritis will be included, in the absence of non-inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Hospitalized in intensive care for management of acute obstructive pyelonephritis
* Patients affiliated to a Social Security System

Exclusion Criteria:

* Pregnancy
* Opposition to data use
* Persons under legal protection (curatorship, guardianship), legal safeguards

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients meeting the eligibility criteria over the period 2015-2022 will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be a combined endpoint of death, and/or stage 3 AKI ( KDIGO classification), and/or non-recovery of renal function. | up to 30 days after admission to intensive care

SECONDARY OUTCOMES:
Death | up to 30 days after admission to intensive care
Stage 3 Acute kidney injury (KDIGO classification) | up to 30 days after admission to intensive care
failure to recover renal function | up to 30 days after admission to intensive care .
  defined as creatinine levels greater than 150% of baseline value
the incidence of acute renal failure defined by KDIGO 1 | up to 30 days after admission to intensive care
the incidence of acute renal failure defined by KDIGO 2 and 3 | up to 30 days after admission to intensive care
the incidence of Renal replacement therapy | up to 30 days after admission to intensive care
the incidence of non-recovery of renal fuction | up to 30 days after admission to intensive care
The number of days alive without Renal replacement therapy | up to 30 days after admission to intensive care
The number of days alive without catecholamines | up to 30 days after admission to intensive care
The number of days alive without antibiotics | up to 30 days after admission to intensive care
The number of days alive without | up to 30 days after admission to intensive care
Death rate | up to 30 days after admission to intensive care

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Dr COUTROT, MD, Principal Investigator — Hopital saint Louis-APHP
Locations (1):
- Hospital Saint Louis, Paris, France

REFERENCES:
- [Background] Kakinoki H, Tobu S, Kakinoki Y, Udo K, Uozumi J, Noguchi M. Risk Factors for Uroseptic Shock in Patients with Urolithiasis-Related Acute Pyelonephritis. Urol Int. 2018;100(1):37-42. doi: 10.1159/000481801. Epub 2017 Oct 24. PMID 29065405
- [Background] Liang X, Huang J, Xing M, He L, Zhu X, Weng Y, Guo Q, Zou W. Risk factors and outcomes of urosepsis in patients with calculous pyonephrosis receiving surgical intervention: a single-center retrospective study. BMC Anesthesiol. 2019 May 1;19(1):61. doi: 10.1186/s12871-019-0729-3. PMID 31039739
- [Background] Yamamoto Y, Fujita K, Nakazawa S, Hayashi T, Tanigawa G, Imamura R, Hosomi M, Wada D, Fujimi S, Yamaguchi S. Clinical characteristics and risk factors for septic shock in patients receiving emergency drainage for acute pyelonephritis with upper urinary tract calculi. BMC Urol. 2012 Mar 13;12:4. doi: 10.1186/1471-2490-12-4. PMID 22413829
- [Background] Baboudjian M, Gondran-Tellier B, Di Bisceglie M, Abdallah R, Michel F, Sichez PC, Al-Balushi K, Akiki A, Gaillet S, Delaporte V, Karsenty G, Lechevallier E, Guieu R, Boissier R. The prognostic value of serum procalcitonin in acute obstructive pyelonephritis. World J Urol. 2021 May;39(5):1583-1589. doi: 10.1007/s00345-020-03353-2. Epub 2020 Jul 15. PMID 32671605
- [Background] Lee SH, Choi T, Choi J, Yoo KH. Differences between Risk Factors for Sepsis and Septic Shock in Obstructive Urolithiasis. J Korean Med Sci. 2020 Nov 9;35(43):e359. doi: 10.3346/jkms.2020.35.e359. PMID 33169555
- [Background] Yamamichi F, Shigemura K, Kitagawa K, Fujisawa M. Comparison between non-septic and septic cases in stone-related obstructive acute pyelonephritis and risk factors for septic shock: A multi-center retrospective study. J Infect Chemother. 2018 Nov;24(11):902-906. doi: 10.1016/j.jiac.2018.08.002. Epub 2018 Aug 30. PMID 30174285
- [Background] Tambo M, Okegawa T, Shishido T, Higashihara E, Nutahara K. Predictors of septic shock in obstructive acute pyelonephritis. World J Urol. 2014 Jun;32(3):803-11. doi: 10.1007/s00345-013-1166-4. Epub 2013 Sep 15. PMID 24037335
- [Background] Srougi V, Moscardi PR, Marchini GS, Berjeaut RH, Torricelli FC, Mesquita JLB, Srougi M, Mazzucchi E. Septic Shock Following Surgical Decompression of Obstructing Ureteral Stones: A Prospective Analysis. J Endourol. 2018 May;32(5):446-450. doi: 10.1089/end.2017.0896. Epub 2018 Mar 20. PMID 29439607
- [Background] Kamei J, Sugihara T, Yasunaga H, Matsui H, Sasabuchi Y, Fujimura T, Homma Y, Kume H. Impact of early ureteral drainage on mortality in obstructive pyelonephritis with urolithiasis: an analysis of the Japanese National Database. World J Urol. 2023 May;41(5):1365-1371. doi: 10.1007/s00345-023-04375-2. Epub 2023 Mar 22. PMID 36947175
- [Background] Kellum JA, Zarbock A, Nadim MK. What endpoints should be used for clinical studies in acute kidney injury? Intensive Care Med. 2017 Jun;43(6):901-903. doi: 10.1007/s00134-017-4732-1. Epub 2017 Mar 2. No abstract available. PMID 28255614